CLINICAL TRIAL: NCT05051449
Title: Increasing Retention in Methadone Maintenance Treatment: Feasibility and Preliminary Efficacy of Ketamine for the Treatment of Patients With OUD and Comorbid Depression (OUDCD)
Brief Title: Ketamine for OUD and Comorbid Depression (OUDCD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study funds were exhausted
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Annabelle Belcher, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00096377
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use Disorder; Depressive Disorder
MeSH Terms: conditions — Opioid-Related Disorders; Depressive Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental)
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine will be administered by a nurse in a 2-week treatment phase, during which participants will receive six IV infusions of 0.5 mg/kg (over 40-50 minutes) ketamine three times per week. Infusion days for patients will be on Mondays, Wednesdays, and Fridays, +/- 1 day. Ketamine infusions will take place at the UMB General Clinical Research Center (GCRC). The GCRC nurse will deliver ketamine within a private exam room. The infusions will last 40-50 min, and the participant will be observed by the GCRC clinical staff for 2 hours post-infusion. Vital signs will be monitored throughout the treatment; specifically, blood pressure, pulse ox and heart rate will be checked prior to treatment, q20 minutes during infusion, and q30-60 minutes after infusion for up to three hours.

SUMMARY:
Methadone is a first-line, evidence-based treatment for opioid use disorder (OUD). Unfortunately, retention and adherence in methadone treatment is a major challenge. OUD patients frequently present with co-morbid depression (OUDCD), a risk factor for poor OUD treatment outcomes, overdose, and suicide. The last two decades have seen an exciting and transformational development in the treatment of depression - ketamine. As a safe, rapid-acting anti-depressant deliverable within the context of methadone maintenance treatment, ketamine could feasibly change the landscape of treatment for OUD patients with comorbid depression. This proposal seeks to evaluate implementation outcomes (feasibility and patient acceptance) as well as preliminary efficacy of ketamine on methadone treatment outcomes for OUD patients (n=6) with comorbid depression and depressive symptoms presenting for methadone treatment.

ELIGIBILITY:
Inclusion Criteria

* From NHS prescreen (no contact, Study Day 0): Between the ages of 18 to 65 years old
* From NHS prescreen (no contact, Study Day 0): Daily use of illicit opioids
* From NHS prescreen (no contact, Study Day 0): Fulfillment of DSM-5/ICD-10 criteria for moderate-to-severe opioid or heroin use disorder
* From NHS prescreen (no contact, Study Day 0): Acceptance into methadone maintenance care for treatment of opioid or heroin use disorder
* From screening for study eligibility (Study Contact Day 1): A total of 10 or more points on the PHQ-9
* From screening for study eligibility (Study Contact Day 1): Have had no prior sustained experience/dependence on ketamine or PCP (i.e., must answer "no" to all four questions on the ketamine/PCP screen)

Exclusion Criteria

* From NHS prescreen (no contact, Study Day 0): Patients transferring from another program of opioid agonist treatment
* From NHS prescreen (no contact, Study Day 0): Electrocardiogram (ECG) findings of tachycardia, prior myocardial infarction, myocardial ischemia, or aberrant conduction
* From NHS prescreen (no contact, Study Day 0): Self-report of recent prescribed or illicit benzodiazepine use ("Xannies", or "bars")
* From NHS prescreen (no contact, Study Day 0): Urine screen positive for pregnancy
* From NHS prescreen (no contact, Study Day 0): Stage 2 hypertension, defined by a systolic blood pressure (SBP) > 140 mmHg or a diastolic blood pressure (DBP) > 90 mmHg
* From NHS prescreen (no contact, Study Day 0): Clinically significant abnormal laboratory values, physical exam findings or self-reported medical conditions for which a transient increase in blood pressure could be significantly detrimental (e.g., cardiovascular disease), as determined by the evaluating intake physician
* From NHS prescreen (no contact, Study Day 0): Any clinically significant abnormal findings from intake health and physical examination
* From NHS prescreen (no contact, Study Day 0): Any indication of serious mental illness or psychiatric disorder from the attending's evaluation notes
* From Liver Function Screen (Study Contact Day 2): Baseline alkaline phosphatase > 2.5 times the upper limit of normal
* From Liver Function Screen (Study Contact Day 2): Baseline aspartate aminotransferase > 3 times the upper limit of normal
* From Psychiatric Evaluation (Study Contact Day 2) Current or previous recreational use of ketamine or PCP
* From Psychiatric Evaluation (Study Contact Day 2): Subjects who meet DSM-5 criteria for current bipolar disorder
* From Psychiatric Evaluation (Study Contact Day 2): Past or current presence of psychotic symptoms, or diagnosis of a lifetime psychotic disorder including schizophrenia or schizoaffective disorder
* Subjects who meet DSM-5 criteria for current or history of psychotic spectrum disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: Study Recruitment | One year
  Feasibility will be assessed via participant recruitment: 50% of eligible patients approached will consent to participation in the pilot.
Feasibility: Study Retention | One year
  75% of participants will be retained throughout the duration of ketamine infusion procedures
Patient Acceptability: Acceptability of the Intervention Measure (AIM) | One month
  Acceptance will be assessed via scores on the Acceptability of the Intervention Measure (AIM): Distribution summarized with mean and 95% C.I. Scale values range from 1 to 5 with higher mean values representing greater agreement and/or acceptability.
Patient Acceptability: Engagement | One month
  Engagement will be assessed via dosing records of observed ketamine administration: distribution of percentage of completed infusions per patient.

SECONDARY OUTCOMES:
Patient Treatment Retention | Three months
  One-month (30-day) methadone treatment retention as a binomial (yes/no) variable outcome.
Changes in Psychiatric Diagnosis of Depression | One month
  Assessment of changes in depression (MADRS score) will be made at baseline and on the final study day based on a Minimal Clinically Important Difference (MCID) defined change of 1.9 points
Changes in Depressive Symptoms | One month
  Assessment of changes in symptoms of depression, measured with the Patient Health Questionnaire (PHQ-9) will be made at baseline and on the final study day.

OTHER OUTCOMES:
Self-report of illicit substance use | One month
  Assessment of changes in number of days of substance use from baseline to the last study contact. Drug use is assessed via self-report of past-two-week use of four common substances: opioids (including heroin, fentanyl, and nonprescribed opioids), cocaine, benzodiazepines, and alcohol; "other" is a fifth category. Total days used (out of a possible 14) is recorded.
Subjective Opioid Withdrawal Scale (SOWS) | One monrh
  Assessment of changes in scores on the SOWS from baseline to the last study contact day. SOWS is a 16-item patient self-report instrument to assess common subjective symptoms of craving and withdrawal.
Objective Opioid Withdrawal Scale (OOWS) | One month
  Assessment of changes in scores on the OOWS from baseline to the last study contact day. The OOWS is a 13-item clinical assessment of observable physiological signs of withdrawal.
Craving Assessment | One month
  Assessment of changes in scores on the Craving Assessment from baseline to the last study contact day. This assessment is an adapted one-item visual-analog scale of self-report of craving for drugs.
Pittsburgh Sleep Quality Index (PSQI) | One month
  Assessment of changes in scores on the PSQI from baseline to the last study contact day. The PSQI is a self-rated 19-item questionnaire that assesses sleep quality and disturbances over a one-month time interval. Seven component scores are generated: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for the 7 components yields one global score. Assessment of changes will be based on the global score.
The Short Inventory of Problems-Revised (SIP-R) | One month
  Assessment of changes in scores on the SIP-R from baseline to the last study contact day. The SIP-R is a 15-item self-report assessment of the adverse consequences of substance use.
Generalized Anxiety Disorder 7-item scale (GAD-7) | One month
  Assessment of changes in scores on the GAD-7 from baseline to the last study contact day. The GAD-7 is a 7-item screen designed to identify individuals with probable anxiety. Each item is scored with a score between 0 and 3 (Not at all sure= 0; Several days= 1; Over half the days= 2; Nearly every day= 3), yielding a total between 0 and 21.
Acceptability of the Intervention (AIM) | One month
  Assessment of changes in scores on the AIM from baseline to the last study contact day. An established implementation instrument used widely in clinical research, the AIM is a 4-item Likert-type measure of acceptability of an intervention.
Clinician Administered Dissociative Symptom Scale (CADSS-6) | Two weeks
  Assessment of changes in scores on the CADSS-6 across ketamine infusion days. The CADSS-6 is a 6-item clinician-administered assessment of treatment-emergent dissociation, an adverse event associated with I.V. ketamine; administered 5-10 minutes following cessation of the ketamine infusion on all infusion days
Drug Effects Questionnaire-5 (DEQ-5) | Two weeks
  Assessment of changes in scores on the CADSS-6 across ketamine infusion days. The DEQ is a five-point self-report visual analogue scale-based assessment of two key aspects of an individual's acute, subjective response to the experience of drug consumption: (i) the strength of substance effects and (ii) desirability of substance effects; administered immediately following CADSS-6 administration.
Modified Aldrete | Two weeks
  This assessment determines safe discharge from the hospital following each day of ketamine infusion, and will be administered just prior to release. This 5-point clinical assessment is used as a post-operative tool to determine safe discharge following anesthesia. Scores of 0 to 2 are assigned to each of five domains, which include Activity, Respiration, Circulation, Consciousness and Oxygen Saturation.

CONTACTS AND LOCATIONS:
Overall Officials: Annabelle Belcher, PhD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No